CLINICAL TRIAL: NCT06576661
Title: Evaluation of the LithoVue Elite Ureteroscope With Intra-Renal Pressure Monitoring Technology: Examination of Surgeon Behavior and Post-operative Outcomes
Acronym: ELITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Bristol Whiles, MD, Professor of Urology, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00160851
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Kidney Stone; Nephrolithiasis
Keywords: Intrarenal Pressure; LithoVue Elite
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- URS WITH INTRARENAL PRESSURE MONITORING VISIBLE (Active Comparator): In Arm 1, participants will undergo URS with real-time IRP monitoring visible to surgeons using the LithoVue Elite™. Participants will be scheduled to undergo URS per standard of care. All follow-up visits will be scheduled per standard of care.
  Interventions: Device: INTRARENAL PRESSURE MONITORING VISIBLE
- URS WITHOUT INTRARENAL PRESSURE MONITORING VISIBLE (No Intervention): In Arm 2, participants will undergo URS LithoVue Elite™ without the real-time IRP monitoring information visible to the surgeon. Participants will be scheduled to undergo URS per standard of care. All follow-up visits will be scheduled per standard of care.

INTERVENTIONS:
Device: INTRARENAL PRESSURE MONITORING VISIBLE — In Arm 1, participants will undergo URS with real-time IRP monitoring visible to surgeons using the LithoVue Elite™.
  Arms: URS WITH INTRARENAL PRESSURE MONITORING VISIBLE

SUMMARY:
The goal of this study is to evaluate the influence of real-time intrarenal pressure measurement availability on surgeons' behavior during ureteroscopy while using the ureteroscope LithoVue Elite.

DETAILED DESCRIPTION:
Despite advances in surgical techniques and technology, preventable adverse events still occur in the operating room, with half of them attributed to poor non-technical skills of surgical teams. Therefore, it is essential to observe and measure surgeons' intraoperative non-technical skills and provide structured feedback to improve patient safety. The new LithoVue Elite™ disposable ureteroscope has the potential to impact surgeons' behavior during ureteroscopy, as it enables the measurement of real-time intrarenal pressures. The study is designed to evaluate urologists' behavior during ureteroscopic stone treatment with and without intra-renal pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over 18 years of age
* Undergoing flexible ureteroscopy to address urinary stones located in the proximal ureter or kidney
* Total stone burden over 2 cm

Exclusion Criteria:

1. Undergoing bilateral stone treatment during the same procedure
2. Patients with known genitourinary anatomical abnormalities
3. Uncorrected coagulopathy
4. Patients with urinary diversions
5. Chronic external urinary catheters
6. Women who are pregnant
7. Immunosuppressed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Surgeon behavior as measured by mean Non-Technical Skills for Surgeons (NOTSS) score. | Procedure
  Treating investigators will be evaluated using the modified NOTSS tool during the procedure. The NOTSS is used to measure non-technical skills in the operation room in the following categories; situation awareness, decision making, communication & teamwork, and leadership.

SECONDARY OUTCOMES:
Difference in decision-making domain scores as measured by the Non-Technical Skills for Surgeons (NOTSS) scores | Procedure
  Treating investigators will be evaluated using the modified NOTSS tool during the procedure. The NOTSS is used to measure non-technical skills in the operation room in the following categories; situation awareness, decision making, communication & teamwork, and leadership.
Post-operative infection | 30-days post-operative
  Patient signs and symptoms concerning for a urinary tract infection, along with a positive urine culture
Perioperative patient outcomes as measured by Clavien-Dindo classification system | Up to 30 days
  Intraoperative complications will be categorized based on the Clavien-Dindo classification system
Post-operative pain as measured by Visual analog scale (VAS) | Immediately post-operative and up to 7 days
  The VAS is a valid and reliable method for quantifying pain intensity on a scale of 0 to 10, where 0 represents no pain and 10 represents the most severe pain possible.
Post-operative pain as measured by opioid use | Immediately post-operative and up to 7 days
  Opioid usage will be tracked

CONTACTS AND LOCATIONS:
Overall Officials: Bristol B Whiles, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers SO Jr, Gawande AA, Kwaan M, Puopolo AL, Yoon C, Brennan TA, Studdert DM. Analysis of surgical errors in closed malpractice claims at 4 liability insurers. Surgery. 2006 Jul;140(1):25-33. doi: 10.1016/j.surg.2006.01.008. PMID 16857439
- [Background] Baker GR, Norton PG, Flintoft V, Blais R, Brown A, Cox J, Etchells E, Ghali WA, Hebert P, Majumdar SR, O'Beirne M, Palacios-Derflingher L, Reid RJ, Sheps S, Tamblyn R. The Canadian Adverse Events Study: the incidence of adverse events among hospital patients in Canada. CMAJ. 2004 May 25;170(11):1678-86. doi: 10.1503/cmaj.1040498. PMID 15159366
- [Background] Yule S, Flin R, Paterson-Brown S, Maran N. Non-technical skills for surgeons in the operating room: a review of the literature. Surgery. 2006 Feb;139(2):140-9. doi: 10.1016/j.surg.2005.06.017. PMID 16455321
- [Background] Yule S, Flin R, Paterson-Brown S, Maran N, Rowley D. Development of a rating system for surgeons' non-technical skills. Med Educ. 2006 Nov;40(11):1098-104. doi: 10.1111/j.1365-2929.2006.02610.x. PMID 17054619
- [Background] Brunckhorst O, Volpe A, van der Poel H, Mottrie A, Ahmed K. Training, Simulation, the Learning Curve, and How to Reduce Complications in Urology. Eur Urol Focus. 2016 Apr;2(1):10-18. doi: 10.1016/j.euf.2016.02.004. Epub 2016 Feb 24. PMID 28723441
- [Background] Tokas T, Skolarikos A, Herrmann TRW, Nagele U; Training and Research in Urological Surgery and Technology (T.R.U.S.T.)-Group. Pressure matters 2: intrarenal pressure ranges during upper-tract endourological procedures. World J Urol. 2019 Jan;37(1):133-142. doi: 10.1007/s00345-018-2379-3. Epub 2018 Jun 18. PMID 29915944